CLINICAL TRIAL: NCT01973855
Title: Syndrome of Fever Associated With Bleeding of Chinese and Western Medicine Diagnosis and Treatment of Infectious Diseases Plans and Severe Clinical Treatment Research
Brief Title: Chinese and Western Medicine Treatment of Fever Associated With Bleeding Symptoms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Xinghua Tan, Director of Department of infection area, Guangzhou 8th People's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX10004301-003
Record Dates: First submitted 2013-10-24; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Viral Haemorrhagic Fever; Dengue Fever
MeSH Terms: conditions — Hemorrhagic Fevers, Viral; Dengue | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM and Western Medicine (Experimental): TCM and Western Medicine:First Infectious diseases soup recipe,every time a dose,Two times a day;Ribavirin 10-15mg per kg every time Western Medicine：Ribavirin 10-15mg per kg every time
  Interventions: Drug: Western Medicine; Drug: TCM and Western Medicine
- Western Medicine (Placebo Comparator): Western Medicine：Ribavirin 10-15mg per kg every time
  Interventions: Drug: TCM and Western Medicine

INTERVENTIONS:
Drug: Western Medicine — Physical cooling,Hydrocortisone
  Other Names: Ribavirin,
  Arms: TCM and Western Medicine
Drug: TCM and Western Medicine — Third Infectious diseases soup recipe
  Other Names: Second Infectious diseases soup recipe and Ribavirin

SUMMARY:
To meet eligibility criteria, this study and informed consent of the syndrome of fever associated with bleeding of infectious diseases, severe patients to carry out multicenter, practical randomized controlled clinical research, to compare the curative effect of western medicine, combining Chinese and western medicine treatment, and security, and pathogenesis of TCM and syndrome, severe immune related factor and syndrome type of traditional Chinese medicine, Chinese medicine prescriptions mechanism research.

DETAILED DESCRIPTION:
Randomized method: using large sample, central randomized, parallel comparison of Chinese and western medicine and western medicine group.

ELIGIBILITY:
Inclusion Criteria:

* Viral diseases, such as dengue fever, kidney of hemorrhagic fever, such as xinjiang hemorrhagic fever; Or clinical has fever associated with bleeding as the main performance, and confirmed as the new emergent infectious diseases

Exclusion Criteria:

* Diagnosed with flu, hand, foot and mouth disease, viral hepatitis (except the carrier), liver cirrhosis after hepatitis, AIDS, rabies, encephalitis, polio, measles, German measles, chickenpox, herpes, infectious mononucleosis, infectious atypical pneumonia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Anytime of the clinical trail from 2011.1.1 to 2015.12.30

SECONDARY OUTCOMES:
Safety outcome | From 2012.1 to 2015.12
  With adverse events as the calculation basis

CONTACTS AND LOCATIONS:
Overall Officials: Tan X Hua, Study Director — Guangzhou 8th hospitol
Locations (1):
- Xi 'an eighth people's hospital, XiAn, Shanxi, China